CLINICAL TRIAL: NCT07012096
Title: Efficacy of Counselling for the Prevention of Hypertension Among Slum Dwellers in Dhaka City, Bangladesh
Brief Title: Efficacy of Counselling for the Prevention of Hypertension (ECoPH)
Acronym: ECoPH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh University of Health Sciences (Other)
Collaborators: Bangladesh University of Professionals (Unknown)
Responsible Party: Principal Investigator, Palash Chandra Banik, Associate Professor, Bangladesh University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LS20221832
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Hypertension; Cardiovascular diseases; counseling intervention; urban slums; randomized controlled trial; preventive healthcare; Dhaka; Good Clinical Practices
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (CG) (Active Comparator): CG-1: Leaflet + Dummy counselling CG-2: Mobile SMS + Dummy counselling CG-3: Leaflet + Mobile SMS + Dummy counselling
  Interventions: Behavioral: Leaflets and mhealth education
- Placebo (Placebo Comparator): CG-4: No intervention + Dummy counselling.
  Interventions: Other: Dummy Placebo
- Intervention group (IG) (Experimental): IG-1: Leaflet + Counselling (WHO Brief interventions) IG-2: Mobile SMS + Counselling (WHO Brief interventions) IG-3: Leaflet + Mobile SMS + Counselling (WHO Brief interventions) IG-4: Counselling (WHO Brief interventions)
  Interventions: Behavioral: counseling, leaflet and mhealth education for hypertension

INTERVENTIONS:
Behavioral: counseling, leaflet and mhealth education for hypertension — Investigators will develop 6 leaflets and 24-SMSs containing messages on the burden of hypertension, consequences, and the benefits of preventing of hypertension, and the healthy practices for preventing hypertension, tobacco, physical inactivity, dietary salt intake, inadequate fruits and vegetables, overweight and obesity, and the use of trans fat. It will be written in plain and simple Bengali. Leaflets will be received by CG-1, CG-3, IG-1 and IG-3. 24-SMSs. Face-to-face counselling (approximately 20 min/session). A total of 20 sessions (1 cycle) will be provided. The session will be repeated if the cycle is over.
  Arms: Intervention group (IG)
Behavioral: Leaflets and mhealth education — Participants will receive 6 leaflets containing messages on the burden of hypertension, consequences, and benefits of prevention of hypertension, and the healthy practices for preventing hypertension.
  Participants will receive 24 SMSs containing the burden of hypertension, consequences, and benefits of prevention of hypertension, and the healthy practices for preventing hypertension.
  And additionally receive a dummy counselling of 5 to 10 minutes informal discussion with the participants, which will not include any health messages that will be received by the participants of the intervention group.
  Arms: Control group (CG)
Other: Dummy Placebo — Participants will only receive a dummy counselling of 5 to 10 minutes informal discussion with the participants, which will not include any health messages that will be received by the participants of the intervention group.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effectiveness of counseling interventions in promoting positive changes in hypertension markers among adult slum dwellers. The intervention is designed to address modifiable risk factors, such as physical inactivity, obesity, unhealthy dietary practices, tobacco and harmful uses of alcohol within a resource-limited community setting. The main question it aims to answer is:

* Is counseling a more effective intervention for the prevention of hypertension among adult slum dwellers in Dhaka city compared to other interventions?

Participants will:

* provide data related to tobacco use, physical activity, and dietary intake.
* provide a sample for blood pressure measurements. Will receive the WHO Brief Counselling intervention through 20 personalised sessions (each lasting approximately 20 minutes), focusing on lifestyle modifications, including physical activity promotion, balanced nutrition, and hypertension awareness.

DETAILED DESCRIPTION:
This study aims to provide valuable insights into the effectiveness of counseling interventions in improving hypertension-related health outcomes among vulnerable urban populations. By focusing on modifiable risk factors, such as physical activity, dietary behavior, and tobacco use, the study will assess the potential of personalized counseling to reduce obesity, improve lipid profiles, and lower blood pressure. The intervention group will receive leaflet and counseling; and the control group will receive a leaflet only. After randomization, we will perform a baseline assessment. The participants will be allocated using stratified randomization. Allocation coverup will be ensured by performing allocation after completing all baseline assessments. A researcher who will not directly be involved with study delivery will allocate participants in a 1:1 ratio, generating a random sequence.

For both the primary and secondary outcomes, an intent-to-treat (ITT) design will be employed to ensure the robustness of the findings by including all participants, regardless of whether they complete the study or drop out. To address the potential impact of missing data due to dropout, participants will still be invited back for final assessment evaluations, minimizing bias in outcome measurement.

Through rigorous monitoring of primary and secondary outcomes in a double-blinded randomized controlled trial, the findings are expected to contribute to evidence-based public health interventions tailored for slum communities in Dhaka. These insights will guide future programs aimed at reducing the burden of hypertension and associated cardiovascular risks. The study will also highlight the importance of community-level preventive strategies in addressing chronic diseases where access to healthcare is limited. Ultimately, the research can inform scalable public health initiatives, advancing efforts toward equitable healthcare solutions in urban low-income settings

ELIGIBILITY:
Inclusion Criteria: People who are not diagnosed as hypertensive patients are healthy and have no history of diseases and stay in the slum for at least one year.

Exclusion Criteria: People who have the following condition will be excluded:

* kidney disease
* psychiatric illness
* including depression
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals whose self-identified gender on their national identity card is listed as (Male/Female/other) are eligible to participate.
Enrollment: 1700 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
BMI classification (kg/m²) | From enrollment until 18 months
  Body mass index (BMI) will be calculated as weight in kilograms divided by height in meters squared (kg/m²). The participants will be considered as obese and over-weight when BMI ≥ 30kg/m2 and 25-29.9 kg/m2, respectively
Waist circumference (cm) | From enrollment until 18 months
  Central obesity was categorized according to the cut-off value specified by the international Diabetes Federation--- waist circumference 90 cm for men and 80 cm for women or waist-hip ratio>0.90 for men and >0.85 for women.
Waist-to-hip ratio | From enrollment until 18 months
  Waist-to-hip ratio will be calculated as the ratio of waist circumference to hip circumference. Central obesity will be defined as a ratio >0.90 in men and >0.85 in women.
Tobacco use in the past 30 days | From enrollment until 18 months
  Those who have the past 30 days history of smoking or use of smokeless tobacco will be considered as a current tobacco user.
Physical activity level (MET-minutes/week) | From enrollment until 18 months
  As per the WHO STEPS protocol, we were converted all work-related physical activities in metabolic equivalent of task in minutes per day (MET-minute) as follows:
  1 minute in sedentary position = 1 MET-minute
  1 minute in a moderate physical activity = 4 MET-minutes
  1 minute in a vigorous physical activity = 8 MET-minutes
  All MET-minutes were then added together to get the cumulative MET-minutes. As per the cumulative MET-minutes, participants were categorized as less, moderately, and highly active:
  * 600 MET-minutes per week = less active
    * 600-3000 MET-minutes per week = moderately active ≥ 3000 MET-minutes per week = highly active
  The rest of the respondents, those didn't not meet even moderate activities, they were categorized as low activity
Inadequate fruit and/or vegetables intake (servings) | From enrollment until 18 months
  WHO recommendation of fruit and/or vegetable intake <5 servings per day was considered as an inadequate intake. Participants will be asked about the number of days they used to eat fruit and vegetables in a week and the number of servings on those days they eat these. One standard serving size equal to 80 grams.
Dietary salt intake | From enrollment until 18 months
  The added salt consumption will be defined as taking dietary salt during eating a meal.

SECONDARY OUTCOMES:
Systolic Blood pressure (mmHg) | From enrollment until 18 months
  The blood pressure of the respondents will be measured following WHO guideline for blood pressure measurement using WHO-certified automated blood pressure monitor namely OMRON model HEM-7121 made in Japan. Hypertension will be defined as SBP ≥140 mmHg or if the participant is on antihypertensive treatment.
Diastolic blood pressure (mmHg) | From enrollment until 18 months
  The participants will be considered hypertensive when the systolic blood pressure reading was ≥140 mmHg and/or the diastolic blood pressure reading was ≥ 90 mmHg or known case hypertensive or on antihypertensive medication. Raised blood pressure means SBP: ≥ 120 mmHg and /or DBP: ≥ 80 mmHg
Heart rate (beats per minute) | From enrollment until 18 months
  Heart rate refers to the number of times the heart beats per minute (bpm). In this study, heart rate will be measured using a validated automated device (OMRON model HEM-7121) following the standard protocols recommended by the World Health Organization. Participants will be instructed to rest for at least five minutes before the measurement to ensure accuracy. Heart rate readings will be taken at baseline and follow-up intervals to track any significant changes over time, with abnormal heart rates defined as below 60 bpm (bradycardia) or above 100 bpm (tachycardia) in accordance with clinical guidelines.
Lipid profile (mg/dL) | From enrollment until 18 months
  Serum total cholesterol, triglycerides and HDL-cholesterol will be measured by end-point method using Backman Coulter AU-480 automated Biochemistry analyzer. Serum LDL-cholesterol will be calculated using Friedewald formula.
  Dyslipidemia was defined as Total Cholesterol ≥ 200 mg/dl, or Triglycerides ≥150 mg/dl, or Low-density lipoprotein cholesterol (LDL-C) ≥ 130 mg/dl, or HDL-C < 40 mg/dl (for men) and High-density lipoprotein cholesterol (HDL-C) < 50 (for women)
Fasting blood glucose (mg/dL) | From enrollment until 18 months
  Fasting blood sugar levels will be measured from venous samples following an 8-hour fast using the Turbidimetric Immunoinhibition methods using Backman Coulter AU-480.
Diagnosis of Type 2 Diabetes Mellitus | From enrollment until 18 months
  Type 2 diabetes mellitus will be diagnosed if fasting blood glucose is ≥126 mg/dL or if the participant is on antidiabetic medication, following WHO criteria.
High-sensitivity C-reactive protein (hs-CRP) (mg/L) | From enrollment until 18 months
  Hs-CRP will be measured using turbidimetric immunoassay methods with a Beckman Coulter AU-480 automated biochemistry analyzer. Blood samples will be collected from participants after fasting, and Hs-CRP levels will be expressed in milligrams per liter (mg/L). Following clinical standards, values below 1 mg/L indicate low cardiovascular risk, 1-3 mg/L represent moderate risk, and above 3 mg/L indicate high cardiovascular risk
Urine creatinine test (mg/dL) | From enrollment until 18 months
  Following instruction on proper urine preservation, participants were given a 15-20 ml sterile labeled container to collect urine for urine specimens, which were to be stored overnight at room temperature before being collected the following morning. The creatinine level was estimated using the Jaffy method and the Backman Coulter AU-480 automated Biochemistry analyzer was used to measure serum creatinine.
Urinary sodium (Na+) and potassium (K+) estimation (mmol/L) | From enrollment until 18 months
  In this investigation, we employed the Tanaka equation to estimate 24-hour urine Na+, K+, and Na+/K+ ratio. The equation used Japanese data items from the INTERSALT project, which was carried out using a highly standardized technique, to build this equation to estimate 24-hour urine Na+ and K+ excretion. By contrasting 24-hour urine samples with spot urine from the same participants, they were able to create this equation. Additional data utilized to create the equation included the respondents' age, sex, height, weight, and creatinine levels. This was then used to get the 24-hour sodium intake, which was then divided by 17.1 as a conversion factor to determine the predicted salt intake in grams. Using the Backman Coulter AU-480 automated biochemistry analyzer, the ISE method will be used to measure the amount of sodium (Na+) in the urine.
10-year cardiovascular disease (CVD) risk prediction | From enrollment until 18 months
  CVD risk will be estimated using WHO/ISH risk prediction charts (version 2023), incorporating factors like age, sex, blood pressure, smoking status, diabetes, and total cholesterol. Risk will be categorized as very low risk <5%, low risk 5%-<10%, moderate risk 10%-<20%, high risk 20%-<30% and very high risk ≥30%

CONTACTS AND LOCATIONS:
Overall Officials: Palash C. Banik, MPhil in Noncommunicable disea, Principal Investigator — Bangladesh University of Health Sciences
Locations (1):
- Kallyanpur Pora slum, Kalyanpur mahalla, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Data will be available upon valid request to the PI through email